CLINICAL TRIAL: NCT03640949
Title: Vasopressin and Methylprednisolone for In-Hospital Cardiac Arrest - A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Vasopressin and Methylprednisolone for In-Hospital Cardiac Arrest
Acronym: VAM-IHCA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lars Wiuff Andersen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Lars Wiuff Andersen, Associate Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00001; 2017-004773-13 (EudraCT Number)
Record Dates: First submitted 2018-08-19; First posted 2018-08-21 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Heart Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Arginine Vasopressin; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vasopressin and methylprednisolone (Experimental): The study drugs will consist of 40 mg methylprednisolone (Solu-medrol®, Pfizer) and 20 IU of vasopressin (Empressin®, Amomed Pharma GmbH) given as soon as possible after the first dose of adrenaline. Additional doses of vasopressin (20 IU) will be administered after each adrenaline dose for a maximum of four doses (80 IU).
  Interventions: Drug: Vasopressin, Arginine; Drug: Methylprednisolone
- Placebo (Placebo Comparator): The placebo for vasopressin will consist of 1 mL of 9 mg/mL NaCl ("normal saline") from 2 mL ampules identical to the vasopressin ampules. The placebo for methylprednisolone will also consist of 1 mL of 9 mg/mL NaCl.
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Vasopressin, Arginine — 20 IE of vasopressin per dose for a maximum of four doses (80 IU)
  Arms: Vasopressin and methylprednisolone
Drug: Methylprednisolone — 40 mg methylprednisolone once
  Arms: Vasopressin and methylprednisolone
Drug: NaCl — Placebo
  Arms: Placebo

SUMMARY:
This is an investigator-initiated, multicenter, randomized, placebo-controlled, parallel group, double-blind, superiority trial of vasopressin and methylprednisolone during adult in-hospital cardiac arrest. There will be ten enrolling sites in Denmark. 492 adult patients with in-hospital cardiac arrest receiving at least one dose of adrenaline will be enrolled. The primary outcome is return of spontaneous circulation and key secondary outcomes include survival at 30 days and survival at 30 days with a favorable neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

1. In-hospital cardiac arrest
2. Age ≥ 18 years
3. Received at least one dose of adrenaline during cardiopulmonary resuscitation

Exclusion Criteria:

1. Clearly documented "do-not-resuscitate" order prior to the cardiac arrest
2. Prior enrollment in the trial
3. Invasive mechanical circulatory support at the time of the cardiac arrest
4. Known or suspected pregnancy at the time of the cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars W Andersen, MD, MPH, PhD, DMSc, Principal Investigator — Aarhus University Hospital
Locations (10):
- Denmark (10):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Copenhagen University Hospital - Gentofte, Hellerup
  - Copenhagen University Hospital - Herlev, Herlev
  - Horsens Regional Hospital, Horsens
  - Zealand University Hospital - Køge, Køge
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing. Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. Data will be completely anonymized according to Danish law.
  All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data. There will be no predetermined end date for the data sharing.
Supporting Information: Study Protocol, SAP
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator. Authorship of publications emerging from the shared data will follow standard authorship guidelines from the International Committee of Medical Journal Editors and might or might not include authors from the steering committee depending on the nature of their involvement.

REFERENCES:
- [Derived] Andersen LW, Isbye D, Kjaergaard J, Kristensen CM, Darling S, Zwisler ST, Fisker S, Schmidt JC, Kirkegaard H, Grejs AM, Rossau JRG, Larsen JM, Rasmussen BS, Riddersholm S, Iversen K, Schultz M, Nielsen JL, Lofgren B, Lauridsen KG, Solling C, Paelestik K, Kjaergaard AG, Due-Rasmussen D, Folke F, Charlot MG, Jepsen RMHG, Wiberg S, Donnino M, Kurth T, Hoybye M, Sindberg B, Holmberg MJ, Granfeldt A. Effect of Vasopressin and Methylprednisolone vs Placebo on Return of Spontaneous Circulation in Patients With In-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2021 Oct 26;326(16):1586-1594. doi: 10.1001/jama.2021.16628. PMID 34587236
- [Derived] Andersen LW, Sindberg B, Holmberg M, Isbye D, Kjaergaard J, Zwisler ST, Darling S, Larsen JM, Rasmussen BS, Lofgren B, Lauridsen KG, Paelestik KB, Solling C, Kjaergaard AG, Due-Rasmussen D, Folke F, Charlot MG, Iversen K, Schultz M, Wiberg S, Jepsen RMHG, Kurth T, Donnino M, Kirkegaard H, Granfeldt A. Vasopressin and methylprednisolone for in-hospital cardiac arrest - Protocol for a randomized, double-blind, placebo-controlled trial. Resusc Plus. 2021 Jan 30;5:100081. doi: 10.1016/j.resplu.2021.100081. eCollection 2021 Mar. PMID 34223347
- See also: Trial website — https://www.vam-ihca.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vasopressin and Methylprednisolone | Placebo
Started | 237 | 264
Completed | 237 | 264
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vasopressin and Methylprednisolone | Placebo | Total
Number analyzed (Participants) | 237 | 264 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (13) | 70 (12) | 71 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 90 | 179
  Male | 148 | 174 | 322
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Return of Spontaneous Circulation
Description: Return of spontaneous circulation is defined as spontaneous circulation with no further need for chest compressions sustained for at least 20 minutes
Time Frame: During the cardiac arrest, an average of 20 minutes
Measure: Number; unit: participants
Arm/Group | Vasopressin and Methylprednisolone | Placebo
Number analyzed (Participants) | 237 | 264
participants | 100 | 86

2. Secondary Outcome: Number of Participants That Survived 30 Days
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Vasopressin and Methylprednisolone | Placebo
Number analyzed (Participants) | 237 | 264
Participants | 23 | 31

3. Secondary Outcome: Number of Participants With a Favorable Neurological Outcome at 30 Days
Description: A favorable neurological outcome will be defined as a cerebral performance category score of 1 or 2. The cerebral performance category score is a 5-point scale assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes.
Time Frame: At 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Vasopressin and Methylprednisolone | Placebo
Number analyzed (Participants) | 237 | 264
Participants | 18 | 20

4. Other Pre Specified Outcome: Vasopressor-free Days
Description: Vasopressor-free days will be defined as the number of days within the first 7 days after the cardiac arrest where the patient is not receiving vasopressors and is alive.
Time Frame: 7 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Invasive Ventilation-free Days
Description: Invasive ventilation-free days will be defined as the number of days within the first 7 days after the cardiac arrest where the patient is not receiving invasive ventilation and is alive.
Time Frame: 7 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Sequential Organ Failure Assessment (SOFA) Score at 24, 48 and 72 Hours
Description: The SOFA score is a validated and widely used measure of organ failure assessing the respiratory, nervous, cardiovascular, hepatic, coagulation, and renal systems. We will assess both the cardiovascular sub score as well as the overall SOFA score.
Time Frame: 24, 48 and 72 hours
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Hospital Disposition
Description: Hospital disposition (e.g. home, rehabilitation, nursing home, hospice) will be defined at the time of discharge from the initial acute care hospital.
Time Frame: At hospital discharge, up to 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Survival
Time Frame: At 90 days, 180 days, and 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Favorable Neurological Outcome
Description: as for outcome 3
Time Frame: At 90 days, 180 days, and 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Modified Rankin Scale (mRS)
Description: The mRS is a 7-point scale, ranging from 0 (no symptoms) to 6 (dead), assessing the degree of disability and dependence after a neurological injury such as stroke or cardiac arrest. A good outcome will be defined as a mRS of 0 to 3 and a poor outcome as 4 to 6.
Time Frame: At 30 days, 90 days, 180 days, and 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Glasgow Outcome Scale Extended (GOSE)
Description: The GOSE is a 8-point scale that is an extension of the Glasgow Outcomes Scale (which is identical to the CPC, only with inverse scores) where the scores 1, 2 and 3 from the CPC score is divided into two.
Time Frame: At 30 days, 90 days, 180 days, and 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Health-related Quality of Life (EQ-5D-5L)
Description: The EQ-5D-5L is a well-established measure of health-related quality of life that is quantified as a utility (i.e. a measure of quality of life between 0 and 1).
Time Frame: At 30 days, 90 days, 180 days, and 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through hospital admission up to 1 year
Arm/Group | Vasopressin and Methylprednisolone | Placebo
All-Cause Mortality (participants affected / at risk) | 214/237 | 233/264
Serious Adverse Events (participants affected / at risk) | 0/237 | 0/264
Other Adverse Events (participants affected / at risk) | 0/237 | 0/264

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT03640949/Prot_SAP_000.pdf